CLINICAL TRIAL: NCT02770872
Title: The Association of SAA With Apolipoprotein B Affects Cardiovascular Risk
Status: Completed | Type: Observational
Sponsor: Lisa Tannock (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Lisa Tannock, Sponsor/PI, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: TAN-14-002-HAF
Record Dates: First submitted 2015-05-11; First posted 2016-05-12 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Cardiovascular Disease
Keywords: serum amyloid a; lipoprotein; insulin resistance; dyslipidemia
MeSH Terms: conditions — Cardiovascular Diseases; Insulin Resistance; Dyslipidemias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood will be collected, which will contain DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Obese, normal: Approximately 25 subjects aged 50-75 with BMI's between 27-45 kg/m2. Observation of SAA on apoB containing lipoproteins
  Interventions: Other: Observation of SAA on apoB containing lipoproteins
- Obese, MetS: Approximately 25 subjects aged 50-75 with BMI's between 27-45 kg/m2, blood pressure above 135/80, HDL less than 40 mg/dl, triglycerides greater the 150 mg/dl and fasting blood glucose greater than 100 mg/dl but less than 126 mg/dl. Observation of SAA on apoB containing lipoproteins
  Interventions: Other: Observation of SAA on apoB containing lipoproteins
- Obese, diabetic: Approximately 25 subjects aged 50-75 with BMI's between 27-45 kg/m2 and physician diagnosed diabetes mellitis. Observation of SAA on apoB containing lipoproteins
  Interventions: Other: Observation of SAA on apoB containing lipoproteins

INTERVENTIONS:
Other: Observation of SAA on apoB containing lipoproteins — attempting to elicit the conditions by which SAA shifts from apo-A1 containing lipoproteins to apoB containing lipoproteins

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of death in developed nations and a major health issue in Veterans. Despite a number of different treatments, cardiovascular disease remains a major health burden, thus further treatments are needed. Individuals with obesity and/or diabetes are at particularly high risk for cardiovascular disease, and research suggests that elevated levels of serum amyloid A (SAA) may contribute to cardiovascular disease, particularly atherosclerosis. In preliminary studies in both mouse and human the investigators have identified that SAA appears to shift between lipid particles. SAA is mainly found on high density lipoprotein (HDL) particles; however, the investigators have found that in both mice and humans with obesity and/or diabetes SAA is found on low density lipoprotein (LDL) and very low density lipoprotein (VLDL) particles, and the investigators hypothesize that the presence of SAA on LDL or VLDL makes these particles more likely to cause cardiovascular disease. To determine what leads SAA to shift between lipid particles, SAA knockout mice will be injected with HDL containing SAA then blood collected at several time points over 24 hours, and the lipid particles will be isolated to measure SAA. In some experiments the investigators will compare different isoforms of SAA, different types of HDL particles, or induce expression of enzymes likely involved in shifting SAA between particles. To determine if the presence of SAA makes lipid particles bind vascular matrix more strongly, the investigators will collect carotid arteries and compare the extent of lipid particles bound to the vascular matrix in the vessel wall when the particles have or do not have SAA present. If this research confirms this hypothesis then the presence of SAA on LDL or VLDL may 1) be a new marker indicating humans at highest risk for cardiovascular disease and 2) be a new target of therapy to prevent cardiovascular disease.

DETAILED DESCRIPTION:
Clinical burden of CVD: CVD is the leading cause of death in developed nations and the VA population is no exception. Despite decades of research, technical, and pharmacological advances, CVD remains a major public health problem. This is partly due to our impaired ability to identify subjects at greatest risk for CVD events and thus the best candidates for pharmacological risk reducing therapies, and partly due to incomplete use or efficacy of currently available therapies. Epidemiological studies have identified major risk factors for CVD including elevated LDL cholesterol, low HDL cholesterol, hypertension, smoking and diabetes. However, despite targeting individuals with these risk factors with aggressive pharmacological interventions, CVD remains a major public health problem. Furthermore, even in individuals with risk factors who are treated with pharmacological or lifestyle interventions the CVD event rates are higher than in those who never had the risk factors. Recent epidemiologic data evaluating the American Heart Association-identified cardiovascular health metrics reported that the prevalence of having CVD risk factors at ideal levels is < 2%10; implying that >98% of the population are candidates for risk reduction. Clearly, health systems cannot cope with pharmacological interventions for such enormous target populations. Thus, additional risk stratifying markers are needed to identify those at highest risk for events and thus at greatest likelihood of benefit. Several biomarkers, including the acute phase reactants C reactive protein (CRP) and serum amyloid A (SAA) have been studied for their role in predicting CVD events. Both CRP and SAA are chronically elevated in individuals with obesity, metabolic syndrome (MetS), diabetes, rheumatoid arthritis, lupus and other chronic inflammatory conditions associated with increased CVD rates, raising the question of whether these biomarkers merely reflect underlying risk or play a causative role in CVD. Although emerging evidence has cast doubt on the role of CRP as a causative factor the investigators and others recently demonstrated that SAA is directly atherogenic in animal models. Thus, in addition to its role as a biomarker for CVD, SAA may play a causal role in CVD.

SAA: SAA is a family of acute phase proteins synthesized primarily in the liver. In healthy individuals SAA concentrations are < 5 mg/L but during an acute phase response SAA can increase up to 1000 mg/L for a few days, then it rapidly returns to baseline levels. However, chronic inflammatory states such as obesity, MetS, diabetes, rheumatoid arthritis etc, are associated with persistently and significantly elevated SAA concentrations of 30-100 mg/L. Acute elevations in SAA are proposed to play a major role in response to injury and inflammation, participating in cholesterol delivery to injured tissues, recruitment of inflammatory cells, and induction of tissue repair cytokines. However, the chronic elevations of SAA now prevalent in modern society likely reflect a maladaptive response and numerous studies are now examining potential roles of SAA in disease pathology. Using murine models in which acute phase SAA is over-expressed, the investigators and others demonstrated direct increases in atherosclerosis development.

SAA and apolipoprotein B (apoB) containing lipoproteins: SAA is a lipid binding apolipoprotein and lipid-free SAA has not been found in vivo. The dogma is that SAA is exclusively an HDL associated lipoprotein; however, the investigators and others have reported SAA on apoB-containing lipoproteins in both mice and humans. Several studies have reported on a complex termed SAA-LDL associated with components of MetS, remnant like particle cholesterol, smoking status, lifestyle interventions, and statin treatment. These studies suggest that SAA-LDL is a risk factor for CVD. In new preliminary studies the investigators demonstrate that SAA has a differential lipoprotein association in diabetes, and in post-prandial lipoprotein metabolism, and the investigators demonstrate that the presence of SAA on apoB-lipoproteins augments their proteoglycan binding, a key step in atherosclerosis development. Thus, emerging evidence suggests that the presence of SAA on apoB-lipoproteins may be a novel CVD risk factor, play a causal role in atherosclerosis, and thus be a therapeutic target.

Post-prandial apoB-lipoprotein metabolism: The various lipoproteins are defined based on size and density criteria, as well as by their protein constituents. However, even within each lipoprotein class there is considerable heterogeneity, as the particles undergo continuous remodeling. Briefly, lipids consumed in the diet associate with apoB-48 to form chylomicrons, which are transported in intestinal lymphatics before entering the bloodstream. Various enzymes act on newly formed chylomicrons shifting lipids and proteins between chylomicrons and HDLs before the chylomicron remnants are taken up by the liver. The liver re-packages the lipids into VLDL particles containing apoB-100. The hydrolysis of VLDL results in smaller apoB-100 particles called VLDL remnants or intermediate density lipoproteins (IDLs). Collectively, these particles are termed triglyceride rich lipoproteins (TGRLs).

Ongoing remodeling of TGRLs by various lipases leads to the formation of LDL. LDL can be taken up by peripheral tissues, including the vasculature, or by the liver. The sub-endothelial retention of apoB-containing particles initiates atherosclerosis.

Post-prandial lipoproteins and CVD: Elevated levels of LDL cholesterol and low levels of HDL cholesterol are documented risk factors for CVD and contribute causally to atherogenesis. However, individuals with obesity, MetS and diabetes do not typically have elevated LDL cholesterol; their dyslipidemia is characterized by elevated triglycerides and low HDL cholesterol. The role of triglycerides as a CVD risk factor remains controversial; however, post-prandial triglycerides may be a more significant risk factor than fasting triglycerides. As humans spend most of their lives in the post-prandial state, there is ongoing interest in the role of post-prandial lipoprotein metabolism in CVD risk. However, most studies have relied on fasting lipoprotein samples; triglycerides are the lipoprotein component most affected by food consumption. The mechanisms accounting for the excess prevalence of CVD in MetS and diabetic subjects beyond that predicted by the traditional CVD risk factors remain unclear; however, insulin resistant states are characterized by increased intestinal apoB48 production, increased TGRL production and delayed lipoprotein clearance, which may contribute to CVD prevalence. Retention of apoB- containing lipoproteins in the vascular wall by the ionic interaction between apoB and proteoglycans, leads to the initiation of atherosclerosis. Lipolysis of VLDL more than doubles its ability to cross the endothelium and deposit lipids in the subendothelial space. TGRLs have proportionately more triglyceride than cholesterol: however, their size means that they can deposit 5-20 times more cholesterol per particle in the subendothelial space compared to an LDL particle. Increased TGRL production and delayed particle clearance increases the likelihood of particle retention and cholesterol deposition in the subendothelial space. The investigators have novel preliminary data demonstrating that the presence of SAA on apoB-containing lipoproteins increases their proteoglycan binding. The investigators propose that the increased presence of SAA on apoB-containing post-prandial lipoproteins in insulin resistant states increases the atherogenicity of these particles and could be a mechanism accounting for the increased CVD prevalence in insulin resistant states such as MetS and diabetes.

HDL metabolism: Like VLDL and LDL, HDL comprises a range of particles; however, HDL does not contain apoB, instead containing apoA-I. HDL is often separated into two major classes by size and density: the large HDL2 and the smaller HDL3. As discussed above, HDL undergoes continuous lipid interchange with various apoB-containing lipoprotein particles. A change in lipoprotein structure or composition by various enzymes is termed remodeling. HDL is typically thought to be an atheroprotective lipoprotein due to its ability to transport cholesterol away from the periphery back to the liver. In addition, HDL has a number of other beneficial properties including anti-inflammatory and anti-oxidative functions. In insulin resistant states HDL levels tend to be low, and some studies suggest its beneficial properties are reduced. Remodeling of lipoproteins affects their functionality and half-life; for example, the remodeling of HDL by CETP (which transfers triglycerides from TGRL to HDL and cholesterol ester from HDL to TGRL) predisposes HDL to enhanced catabolism and is thought to contribute to the lower levels of HDL seen in insulin resistant states. Although the paradigm is that SAA is a HDL associated lipoprotein, in preliminary studies the investigators have found SAA on apoB particles in insulin resistant persons in the post-prandial period. However, it is not clear how SAA associates with either HDL or apoB-lipoprotein particles.

SAA lipoprotein association: In the setting of an acute phase response SAA levels can increase up to 1000-fold; however, even at these highly elevated levels SAA remains exclusively found on HDL particles. Thus, there is no evidence of a "maximum capacity" of HDL for SAA. How SAA associates with either HDL or apoB-lipoprotein particles is not fully understood. SAA is thought to be produced by the liver in a lipid-free form and bind lipoproteins extracellularly, or in plasma SAA has been shown to induce HDL biogenesis via ATP binding cassette 1 (ABCA1), which may be a major mechanism by which SAA associates with HDL. Murine studies using knockout mice demonstrated that in the absence of HDL, SAA was found on apoB-particles. However, the investigators and others have reported SAA on apoB particles despite the presence of HDL. In new preliminary studies the investigators found that the remodeling of HDL led to the liberation of both lipid-poor apoA-I and lipid-poor SAA, and that lipid-poor SAA associates with apoB particles. Thus, the remodeling of HDL, particularly in the post-prandial period, may lead to SAA shifting from HDL to apoB particles; alternately, SAA could associate with apoB particles during their hepatic secretion. Both HDL remodeling and hepatic apoB- particle secretion are increased in insulin resistant conditions.

Role of lipoprotein-proteoglycan interactions in atherogenesis: There are several hypotheses as to what triggers the initiation of atherosclerosis, with the "Response to Retention" hypothesis well supported by biomedical evidence. As outlined in this theory, early fatty streak lesions are initiated by deposition of atherogenic lipoproteins (LDLs and TGRLs) in the subendothelial matrix by their retention by extra cellular matrix proteoglycans. Studies show that lipoproteins migrate in and out of the subendothelial space, but once bound to proteoglycans these lipoproteins are retained in this region, become more susceptible to oxidation and other modifications, and are taken up by macrophages leading to the formation of foam cells. TGRLs may be even more atherogenic than LDLs as they don't need modification to be taken up by macrophages, and deliver 5-20 times more cholesterol than LDL on per particle basis. The investigators have demonstrated the presence of SAA on apoB-containing lipoprotein particles in mice, and recently confirmed this in humans. In preliminary studies the investigators demonstrate that the presence of SAA on apoB-lipoproteins enhances their proteoglycan binding. The investigators propose that the presence of SAA on apoB-containing lipoproteins enhances their retention increasing atherogenesis.

ELIGIBILITY:
Inclusion Criteria:

Up to 80 U.S. veterans age 50-75 will be recruited in the following three groups:

* Obese (BMI 27-45 kg/m2), metabolically healthy, (25-30 subjects)
* Obese (BMI 27-45 kg/m2), metabolic syndrome, (25-30 subjects)
* Obese (BMI 27-45 kg/m2), diabetic, (25-30 subjects)

Exclusion Criteria:

The use of:

* Statins (we will not exclude subjects on lipid lowering medications if they are willing to discontinue them for 1-2 weeks prior to participation)
* Fibrates
* Niacin
* Anti-inflammatory drugs including Thiazolidinediones, non-steroidal anti-inflammatories (NSAID), aspirin, steroids
* Estrogen replacement

Conditions such as:

* Acute illness
* Chronic inflammatory illness (such as psoriasis, rheumatoid arthritis, lupus, etc.)
* Infections
* Impaired renal function (eGFR < 60 ml/min)
* Hypo- or hyperthyroidism (subjects biochemically euthyroid on levothyroxine therapy are permitted)
* Gastrointestinal dysfunction

Lifestyles including:

* Use of tobacco products
* Consumption of > 3 drinks /day

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will recruit male and female subjects eligible for medical care within the VA healthcare system
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2014-02; Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Post-prandial SAA content on apoB containing lipoproteins after consumption of a high fat shake | Baseline and once every hour for 8 hours. Study completed in a single day
  Subjects will arrive at the clinic fasted and have an IV line established. A baseline blood sample will be drawn at hour zero. The subject will then consume a high fat shake within a 15 minute window. Blood samples will then be drawn every hour for eight hours to determine the time course of SAA shifting from HDL to apoB containing lipoproteins.
Degree of insulin resistance | 4.5 hour study completed in a single day
  Subjects will arrive at the clinic fasted. The subject will have IV sites established in both arms and two baseline blood samples will be drawn (-30 and -10 minute). At time zero, a bolus of glucose will be injected followed by blood sample collection. Blood will be collected at the following time points in minutes; 0, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 19. At time 20 minutes, the subject will receive an IV bolus of insulin and frequent blood sampling will continue at the following time points in minutes; 20, 22, 23, 24, 25, 27, 30, 40, 50, 70, 90, 100, 120, 140 ,160, 180, 210, 240. A total of 32 blood samples will be collected over the course of 4.5 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa R Tannock, MD, Principal Investigator — VA Medical System
Locations (1):
- VA Medical Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Williams KJ, Tabas I. The response-to-retention hypothesis of early atherogenesis. Arterioscler Thromb Vasc Biol. 1995 May;15(5):551-61. doi: 10.1161/01.atv.15.5.551. No abstract available. PMID 7749869
- [Background] Dong Z, Wu T, Qin W, An C, Wang Z, Zhang M, Zhang Y, Zhang C, An F. Serum amyloid A directly accelerates the progression of atherosclerosis in apolipoprotein E-deficient mice. Mol Med. 2011;17(11-12):1357-64. doi: 10.2119/molmed.2011.00186. Epub 2011 Sep 21. PMID 21953420
- [Background] Yang Q, Cogswell ME, Flanders WD, Hong Y, Zhang Z, Loustalot F, Gillespie C, Merritt R, Hu FB. Trends in cardiovascular health metrics and associations with all-cause and CVD mortality among US adults. JAMA. 2012 Mar 28;307(12):1273-83. doi: 10.1001/jama.2012.339. Epub 2012 Mar 16. PMID 22427615
- [Background] Genest J. C-reactive protein: risk factor, biomarker and/or therapeutic target? Can J Cardiol. 2010 Mar;26 Suppl A:41A-44A. doi: 10.1016/s0828-282x(10)71061-8. PMID 20386760
- [Background] Kisilevsky R, Manley PN. Acute-phase serum amyloid A: perspectives on its physiological and pathological roles. Amyloid. 2012 Mar;19(1):5-14. doi: 10.3109/13506129.2011.654294. Epub 2012 Feb 10. PMID 22320226
- [Background] Kotani K, Satoh N, Kato Y, Araki R, Koyama K, Okajima T, Tanabe M, Oishi M, Yamakage H, Yamada K, Hattori M, Shimatsu A; Japan Obesity and Metabolic Syndrome Study Group. A novel oxidized low-density lipoprotein marker, serum amyloid A-LDL, is associated with obesity and the metabolic syndrome. Atherosclerosis. 2009 Jun;204(2):526-31. doi: 10.1016/j.atherosclerosis.2008.09.017. Epub 2008 Sep 27. PMID 19007930
- [Background] Kotani K, Asahara-Satoh N, Kato Y, Araki R, Himeno A, Yamakage H, Koyama K, Tanabe M, Oishi M, Okajima T, Shimatsu A; Japan Obesity and Metabolic Syndrome Study (JOMS) Group. Remnant-like particle cholesterol and serum amyloid A-low-density lipoprotein levels in obese subjects with metabolic syndrome. J Clin Lipidol. 2011 Sep-Oct;5(5):395-400. doi: 10.1016/j.jacl.2011.08.001. Epub 2011 Aug 12. PMID 21981841
- [Background] Kotani K, Satoh-Asahara N, Kato Y, Araki R, Himeno A, Yamakage H, Koyama K, Tanabe M, Oishi M, Okajima T, Shimatsu A; Japan Obesity and Metabolic Syndrome Study Group. Serum amyloid A low-density lipoprotein levels and smoking status in obese Japanese patients. J Int Med Res. 2011;39(5):1917-22. doi: 10.1177/147323001103900536. PMID 22117994
- [Background] Kotani K, Koibuchi H, Yamada T, Taniguchi N. The effects of lifestyle modification on a new oxidized low-density lipoprotein marker, serum amyloid A-LDL, in subjects with primary lipid disorder. Clin Chim Acta. 2009 Nov;409(1-2):67-9. doi: 10.1016/j.cca.2009.08.019. Epub 2009 Aug 29. PMID 19723514
- [Background] Kotani K, Yamada T, Miyamoto M, Ishibashi S, Taniguchi N, Gugliucci A. Influence of atorvastatin on serum amyloid A-low density lipoprotein complex in hypercholesterolemic patients. Pharmacol Rep. 2012;64(1):212-6. doi: 10.1016/s1734-1140(12)70748-x. PMID 22580538
- [Background] Bansal S, Buring JE, Rifai N, Mora S, Sacks FM, Ridker PM. Fasting compared with nonfasting triglycerides and risk of cardiovascular events in women. JAMA. 2007 Jul 18;298(3):309-16. doi: 10.1001/jama.298.3.309. PMID 17635891
- [Background] Lindman AS, Veierod MB, Tverdal A, Pedersen JI, Selmer R. Nonfasting triglycerides and risk of cardiovascular death in men and women from the Norwegian Counties Study. Eur J Epidemiol. 2010 Nov;25(11):789-98. doi: 10.1007/s10654-010-9501-1. Epub 2010 Oct 2. PMID 20890636
- [Background] Nordestgaard BG, Benn M, Schnohr P, Tybjaerg-Hansen A. Nonfasting triglycerides and risk of myocardial infarction, ischemic heart disease, and death in men and women. JAMA. 2007 Jul 18;298(3):299-308. doi: 10.1001/jama.298.3.299. PMID 17635890
- [Background] Pang J, Chan DC, Barrett PH, Watts GF. Postprandial dyslipidaemia and diabetes: mechanistic and therapeutic aspects. Curr Opin Lipidol. 2012 Aug;23(4):303-9. doi: 10.1097/MOL.0b013e328354c790. PMID 22595742
- [Background] Rutledge JC, Mullick AE, Gardner G, Goldberg IJ. Direct visualization of lipid deposition and reverse lipid transport in a perfused artery : roles of VLDL and HDL. Circ Res. 2000 Apr 14;86(7):768-73. doi: 10.1161/01.res.86.7.768. PMID 10764410
- [Background] Lamarche B, Uffelman KD, Carpentier A, Cohn JS, Steiner G, Barrett PH, Lewis GF. Triglyceride enrichment of HDL enhances in vivo metabolic clearance of HDL apo A-I in healthy men. J Clin Invest. 1999 Apr;103(8):1191-9. doi: 10.1172/JCI5286. PMID 10207171
- [Background] Rashid S, Watanabe T, Sakaue T, Lewis GF. Mechanisms of HDL lowering in insulin resistant, hypertriglyceridemic states: the combined effect of HDL triglyceride enrichment and elevated hepatic lipase activity. Clin Biochem. 2003 Sep;36(6):421-9. doi: 10.1016/s0009-9120(03)00078-x. PMID 12951168
- [Background] Hoffman JS, Benditt EP. Secretion of serum amyloid protein and assembly of serum amyloid protein-rich high density lipoprotein in primary mouse hepatocyte culture. J Biol Chem. 1982 Sep 10;257(17):10518-22. PMID 6809750
- [Background] Hu W, Abe-Dohmae S, Tsujita M, Iwamoto N, Ogikubo O, Otsuka T, Kumon Y, Yokoyama S. Biogenesis of HDL by SAA is dependent on ABCA1 in the liver in vivo. J Lipid Res. 2008 Feb;49(2):386-93. doi: 10.1194/jlr.M700402-JLR200. Epub 2007 Nov 21. PMID 18033752
- [Background] Cabana VG, Feng N, Reardon CA, Lukens J, Webb NR, de Beer FC, Getz GS. Influence of apoA-I and apoE on the formation of serum amyloid A-containing lipoproteins in vivo and in vitro. J Lipid Res. 2004 Feb;45(2):317-25. doi: 10.1194/jlr.M300414-JLR200. Epub 2003 Nov 1. PMID 14595002
- [Background] Tamminen M, Mottino G, Qiao JH, Breslow JL, Frank JS. Ultrastructure of early lipid accumulation in ApoE-deficient mice. Arterioscler Thromb Vasc Biol. 1999 Apr;19(4):847-53. doi: 10.1161/01.atv.19.4.847. PMID 10195908
- [Background] Camejo G, Hurt E, Wiklund O, Rosengren B, Lopez F, Bondjers G. Modifications of low-density lipoprotein induced by arterial proteoglycans and chondroitin-6-sulfate. Biochim Biophys Acta. 1991 Apr 15;1096(3):253-61. doi: 10.1016/0925-4439(91)90013-y. PMID 2018799
- [Background] Hurt-Camejo E, Camejo G, Rosengren B, Lopez F, Ahlstrom C, Fager G, Bondjers G. Effect of arterial proteoglycans and glycosaminoglycans on low density lipoprotein oxidation and its uptake by human macrophages and arterial smooth muscle cells. Arterioscler Thromb. 1992 May;12(5):569-83. doi: 10.1161/01.atv.12.5.569. PMID 1576119
- [Background] Schwenke DC, Carew TE. Initiation of atherosclerotic lesions in cholesterol-fed rabbits. II. Selective retention of LDL vs. selective increases in LDL permeability in susceptible sites of arteries. Arteriosclerosis. 1989 Nov-Dec;9(6):908-18. doi: 10.1161/01.atv.9.6.908. PMID 2590068
- [Background] Schwenke DC, Carew TE. Initiation of atherosclerotic lesions in cholesterol-fed rabbits. I. Focal increases in arterial LDL concentration precede development of fatty streak lesions. Arteriosclerosis. 1989 Nov-Dec;9(6):895-907. doi: 10.1161/01.atv.9.6.895. PMID 2590067
- [Background] Schwartz EA, Reaven PD. Lipolysis of triglyceride-rich lipoproteins, vascular inflammation, and atherosclerosis. Biochim Biophys Acta. 2012 May;1821(5):858-66. doi: 10.1016/j.bbalip.2011.09.021. Epub 2011 Oct 7. PMID 22001233
- [Background] Skalen K, Gustafsson M, Rydberg EK, Hulten LM, Wiklund O, Innerarity TL, Boren J. Subendothelial retention of atherogenic lipoproteins in early atherosclerosis. Nature. 2002 Jun 13;417(6890):750-4. doi: 10.1038/nature00804. PMID 12066187
- [Background] Gustafsson M, Levin M, Skalen K, Perman J, Friden V, Jirholt P, Olofsson SO, Fazio S, Linton MF, Semenkovich CF, Olivecrona G, Boren J. Retention of low-density lipoprotein in atherosclerotic lesions of the mouse: evidence for a role of lipoprotein lipase. Circ Res. 2007 Oct 12;101(8):777-83. doi: 10.1161/CIRCRESAHA.107.149666. Epub 2007 Aug 30. PMID 17761930
- [Background] Chiba T, Chang MY, Wang S, Wight TN, McMillen TS, Oram JF, Vaisar T, Heinecke JW, De Beer FC, De Beer MC, Chait A. Serum amyloid A facilitates the binding of high-density lipoprotein from mice injected with lipopolysaccharide to vascular proteoglycans. Arterioscler Thromb Vasc Biol. 2011 Jun;31(6):1326-32. doi: 10.1161/ATVBAHA.111.226159. Epub 2011 Apr 7. PMID 21474830
- [Background] O'Brien KD, McDonald TO, Kunjathoor V, Eng K, Knopp EA, Lewis K, Lopez R, Kirk EA, Chait A, Wight TN, deBeer FC, LeBoeuf RC. Serum amyloid A and lipoprotein retention in murine models of atherosclerosis. Arterioscler Thromb Vasc Biol. 2005 Apr;25(4):785-90. doi: 10.1161/01.ATV.0000158383.65277.2b. Epub 2005 Feb 3. PMID 15692094